CLINICAL TRIAL: NCT02443532
Title: Quality of Life, Treatment Satisfaction, Fear of Hypoglycemia, Eating Habits, Ang Glucose Control in Patients With Type 1 Diabetes: Effects of Structured Group Education Versus Group Care.
Brief Title: Effects of Structured Group Education on Quality of Life and Glycemic Control in Type 1 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Edoardo Mannucci, Director, Diabetology Unit, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIAB120001
Record Dates: First submitted 2015-05-04; First posted 2015-05-14 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured Group education (Experimental): Six weekly interactive group sessions of 4 hours each, providing information and developing skills for diabetes self-management, including eating habits, food composition, calculation of bolus insulin, information on physical exercise, blood glucose self-monitoring, management of hypoglycemia.
  Interventions: Behavioral: Structured group education
- Individual education (Other): Usual care (individual consultations as routinely performed)
  Interventions: Behavioral: Individual education

INTERVENTIONS:
Behavioral: Structured group education — The group intervention consists of interactive sessions for groups of 5-7 patients, dealing with different aspects of management of type 1 diabetes: insulin therapy and hypoglycemia, management of insulin doses, diet, physical exercise, sick days, etc. The intervention is designed for the acquisition of specific skills of self-management. This intervention is provided by a team including physicians, dietitians, and nurses.
  Arms: Structured Group education
Behavioral: Individual education — Usual care (individual consultations as routinely performed)
  Arms: Individual education

SUMMARY:
Patients with type 1 diabetes aged 15-65 years without major complications will be randomized either to usual care or to a structured group education program, with 6 four-hour weekly interactive sessions devoted to diabetes management. The principal endpoint will be the variation of HbA1c at 12 months from enrolment. Secondary endpoints will include quality of life, treatment satisfaction, fear of hypoglycemia, incidence of hypoglycemia.

DETAILED DESCRIPTION:
The group intervention consists of interactive sessions for groups of 5-7 patients, dealing with different aspects of management of type 1 diabetes: insulin therapy and hypoglycemia, management of insulin doses, diet, physical exercise, sick days, etc. The intervention is designed for the acquisition of specific skills of self-management. This intervention is provided by a team including physicians, dietitians, and nurses.

The control group will receive individual education during routine clinic visits, following usual care, complying with the recommendations of national (Italian) guidelines.

HbA1c will be assessed every three months for all the duration of the study. The principal endpoint will be variation from baseline of HbA1c at 12 weeks from the beginning of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes

Exclusion Criteria:

* serious diabetic complications, such as to interfere with physical functioning (e.g., lower limb amputation, renal failure requiring dialysis, blindness)
* Illiteracy

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-03; Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
HbA1c (between-group difference in variation from baseline) | 12 months

SECONDARY OUTCOMES:
Quality of life (Well-being enquiry in Diabetics [WED] questionnaire) | 12 months
Treatment satisfaction (Diabetes Treatment Satisfaction [DTS] questionnaire) | 12 months
Fear of hypoglycemia (Fear of Hypoglycemia [FH-15] questionnaire) | 12 months
Severe hypoglycemia (incidence of episodes of hypoglycemia requiring hospitalization and/or help from third parties, self-reported) | 12 months